CLINICAL TRIAL: NCT01194908
Title: Phase I/II Trial of Tamoxifen Following Epigenetic Regeneration of Estrogen Receptor Using Decitabine and LBH 589 in Patients With Triple Negative Metastatic Breast Cancer
Brief Title: Re-expression of ER in Triple Negative Breast Cancers
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Emory University (Other)
Collaborators: Novartis (Industry); Eisai Inc. (Industry)
Responsible Party: Principal Investigator, Ruth O'Regan, Physician, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00029718; WCI1696-09 (Other: Other)
Record Dates: First submitted 2010-09-01; First posted 2010-09-03 (Estimated); Results first posted 2015-01-26 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Breast Cancer; Breast Tumors; Breast Neoplasms
Keywords: Breast Cancer; Breast Tumors; Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — Decitabine; Panobinostat; Tamoxifen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm A (Experimental): Patients treated with decitabine and LBH589
  Interventions: Drug: Decitabine, LBH589, Tamoxifen

INTERVENTIONS:
Drug: Decitabine, LBH589, Tamoxifen — Dose level -1; Decitabine (IV)(D1-5): 5mg/m2; LBH589 (IV)(D1,8): 10mg/m2
  Dose level 0; Decitabine (IV)(D1-5): 10mg/m2; LBH589 (IV)(D1,8): 10mg/m2
  Dose level +1; Decitabine (IV)(D1-5): 10mg/m2; LBH589 (IV)(D1,8): 15mg/m2
  Dose level +2; Decitabine (IV)(D1-5): 10mg/m2; LBH589 (IV)(D1,8): 20mg/m2
  Dose level +3; Decitabine (IV)(D1-5): 15mg/m2; LBH589 (IV)(D1,8): 20mg/m2
  Dose level +4; Decitabine (IV)(D1-5): 20mg/m2; LBH589 (IV)(D1,8): 20mg/m2
  Other Names: LBH589; Decitabine; Dacogen; Novaldex

SUMMARY:
Patients are being asked to take part in this study because they have metastatic breast cancer that is triple negative (does not express estrogen receptor (ER), progesterone receptor (PR) or HER2). This means that agents such as trastuzumab (Herceptin®) and tamoxifen are not currently treatment options for their cancer. Another option for treating the patient's cancer at this point is with chemotherapy. The patient should discuss this and other options with their doctor prior to entering this study.

Laboratory studies have demonstrated that ER is actually present in some triple negative breast cancers but is "silenced" (does not function properly) because methyl and histone groups are attached to it and inactivate it. Special drugs called demethylating inhibitors (such as decitabine) and histone deacetylase inhibitors (such as LBH589) can remove these methyl and histone groups and reactivate ER. This reactivated ER can then be targeted with agents like tamoxifen.

The patient is being asked to join this clinical research study to find out if ER can be reactivated in their cancer using decitabine in combination with LBH589. If ER is reactivated in their cancer, we will then determine if tamoxifen can decrease the growth of the cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed triple negative (ER-, PR-, HER2-) metastatic or locally advanced breast cancer
* Measurable disease according to the Response Evaluation Criteria in Solid Tumors (RECIST) criteria.
* Disease that is assessable to biopsy for hormone receptor measurement
* At least one line of therapy prior to study entry (acceptable therapies include chemotherapy ± anti-angiogenic therapy). Other investigational therapies except DNA methyltransferase (DNMT) and histone deacetylase (HDAC) inhibitors are allowed.
* Age > 18 years
* Eastern Cooperative Oncology Group (ECOG) Performance Score of 0 or 1 (Appendix A)
* Adequate bone marrow as evidenced by:

  * Absolute neutrophil count > 1,500/μL
  * Platelet count > 100,000/μL
* Adequate renal function as evidenced by serum creatinine < 1.5 mg/dL
* Adequate hepatic function as evidenced by:

  * Serum total bilirubin < 1.5 mg/dL
  * Alkaline phosphatase < 3 times the upper limit of normal (ULN) for the reference lab (< 5 times the ULN for patients with known hepatic metastases
  * Serum glutamic-oxaloacetic transaminase (SGOT)/serum glutamic-pyruvic transaminase (SGPT) < 3 times the ULN for the reference lab (< 5 times the ULN for patients with known hepatic metastases
* Patients must be recovered from both the acute and late effects of any prior surgery, radiotherapy or other antineoplastic therapy
* Patients or their legal representatives must be able to read, understand and provide informed consent to participate in the trial.
* Consent to biopsy before and after therapy with decitabine and LBH589.
* Patients of childbearing potential and their partners must agree to use an effective form of contraception during the study and for 90 days following the last dose of study medication (an effective form of contraception is an oral contraceptive or a double barrier method)

Exclusion Criteria:

* Patients with an active infection or with a fever > 101.30 F within 3 days of the first scheduled day of protocol treatment
* Patients with active central nervous system (CNS) metastases. Patients with stable CNS disease, who have undergone radiotherapy at least 4 weeks prior to the planned first protocol treatment and who have been on a stable dose of corticosteroids for >3 weeks are eligible for the trial
* History of prior malignancy within the past 5 years except for curatively treated basal cell carcinoma of the skin, cervical intra-epithelial neoplasia, or localized prostate cancer with a current prostate-specific antigen (PSA) of < 1.0 mg/dL on 2 successive evaluations, at least 3 months apart, with the most recent evaluation no more than 4 weeks prior to entry
* Patients with known hypersensitivity to any of the components of decitabine or LBH589
* Patients who received radiotherapy to more than 25% of their bone marrow; or patients who received any radiotherapy within 4 weeks of entry
* Patients who are receiving concurrent investigational therapy or who have received investigational therapy within 28 days of the first scheduled day of protocol treatment (investigational therapy is defined as treatment for which there is currently no regulatory authority approved indication)
* Peripheral neuropathy >= Grade 2
* Patients who are pregnant or lactating
* Any other medical condition, including mental illness or substance abuse, deemed by the Investigator to be likely to interfere with a patient's ability to sign informed consent, cooperate and participate in the study, or interfere with the interpretation of the results.
* History of allogeneic transplant
* Known HIV or Hepatitis B or C (active, previously treated or both)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2010-07; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ruth O'Regan, MD, Principal Investigator — Emory University Winship Cancer Institute
Locations (1):
- Emory University Winship Cancer Institute, Atlanta, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A: Patients treated with decitabine and LBH589
  Decitabine, LBH589, Tamoxifen: Dose level -1; Decitabine (IV)(D1-5): 5mg/m2; LBH589 (IV)(D1,8): 10mg/m2
  Dose level 0; Decitabine (IV)(D1-5): 10mg/m2; LBH589 (IV)(D1,8): 10mg/m2
  Dose level +1; Decitabine (IV)(D1-5): 10mg/m2; LBH589 (IV)(D1,8): 15mg/m2
  Dose level +2; Decitabine (IV)(D1-5): 10mg/m2; LBH589 (IV)(D1,8): 20mg/m2
  Dose level +3; Decitabine (IV)(D1-5): 15mg/m2; LBH589 (IV)(D1,8): 20mg/m2
  Dose level +4; Decitabine (IV)(D1-5): 20mg/m2; LBH589 (IV)(D1,8): 20mg/m2
Period: Overall Study
Arm/Group | Arm A
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Arm A
Number analyzed (Participants) | 5
Age, Customized [Number; unit: participants]
  30-39 years | 1
  40-49 years | 2
  50-59 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: To Determine the Maximum Tolerated Dose of Decitabine and LBH589 Given in Combination in Patients With Metastatic or Locally Advanced Metastatic Breast Cancers
Time Frame: Estrogen receptor status checked 5 days after treatment. Staging is done every 8 weeks.
Population: No data were analyzed due to trial termination.
Arm/Group | Arm A
Number analyzed (Participants) | 0

2. Secondary Outcome: To Determine the Safety of Tamoxifen in Combination With Decitabine and LBH589
Time Frame: Patients will undergo an evaluation for extent of disease 8 weeks from starting study drugs and every 8 weeks (2 cycles) while on study.
Population: No data were analyzed due to trial termination.
Arm/Group | Arm A
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Arm A
Serious Adverse Events (participants affected / at risk) | 4/5
Other Adverse Events (participants affected / at risk) | 0/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (N=5)
Death (General disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes